CLINICAL TRIAL: NCT05397340
Title: Deep Brain Stimulation of Asymmetric Targets Versus Bilateral Subthalamic Nucleus (STN) for Parkinson's Disease With Postural Instability/Gait Difficulty: a Prospective, Randomized, Double-blinded Trial
Brief Title: Asymmetric Targeted DBS for PD With PIGD
Acronym: ATS-PIGD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Asym Stim-PIGD
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: postural instability/gait difficulty; deep brain stimulation; subthalamic nucleus; globus pallidus internus
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-GPi/R-STN (Experimental): Participants randomized in this arm will receive L-GPi/R-STN stimulation for 1 year.
  Interventions: Device: Deep brain stimulation
- Bi-STN (Active Comparator): Participants randomized in this arm will receive bilateral STN stimulation for 1 year.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — active DBS with optimal stimulating parameters

SUMMARY:
The purpose of this study is to compare the effectiveness of the deep brain stimulation of asymmetric targets [subthalamic nucleus (STN) in the right hemisphere while globus pallidus interna (GPi) in the left] versus the bilateral STN for the treatment of Parkinson's disease (PD) with postural instability/gait difficulty (PIGD) in a randomized, double-blinded manner.

DETAILED DESCRIPTION:
This is a double-blinded, randomized, controlled trial aiming at comparing the efficacy of asymmetric targets and bilateral STN DBS in treating PD with PIGD.

After being informed about the study and potential risks, enrolled patients giving written informed consent will be screened to determine eligibility for study entry. Patients who meet the eligibility requirements will be randomized into two groups in a 1:1 ratio using a minimization randomization method in a double-blinded manner, and later undergo bilateral DBS surgery. One group of patients will receive stimulation of left GPi and right STN, while the other will receive STN stimulation bilaterally. The follow-up period will be one year, with corresponding clinical assessments completed at six months and one year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease
* postural instability/gait difficulty (PIGD) phenotypes in the on-medication condition

Exclusion Criteria:

* Atypical parkinsonism
* History of stroke, encephalitis, neuroleptic uses, MRI scan with evidence of significant brain atrophy, lacunar infracts, or other conditions that might interfere with intracranial surgery
* Presence of cognitive, or psychiatric or other co-morbidities (e.g., dementia, epilepsy, cranial traumatism, brain tumor, schizophrenia, severe depression or bipolar disorder, personality disorder, etc.) that might interfere with the patient's ability to complete the evaluations or to provide informed consent
* Presence of anatomical abnormalities in the target region
* Clinically significant medical history that would increase pre-/post-operative complications
* Other conditions considered by the investigators that might interfere with the surgery procedure, the follow-ups, and the interpretation of the data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Movement Disorder Society-sponsord Unified Parkinson's Disease Rating Scale Part III at 12 months | Baseline and 12 months
  In the off-medication condition, scores could range from 0 (no movement symptoms) to 72 (severe movement symptoms).
Change from Baseline in balance ability on the Burg Balance Scale (BBS) at 12 months | Baseline and 12 months
  In the off-medication condition, the scores could range from 0 (severe balance problem) to 56 (no balance problem).
Change from Baseline in the number of freezing episodes on the Timed Up and Go test at 12 months | Baseline and 12 months
  in the off-medication condition

SECONDARY OUTCOMES:
Change from Baseline in completion time on the Timed Up and Go test at 12 months | Baseline and 12 months
  in the off-medication condition
Change from Baseline in completion time on the Timed Up and Go test at 6 months | Baseline and 6 months
  in the off-medication condition
Change from Baseline in the number of steps on the Timed Up and Go test at 12 months | Baseline and 12 months
  in the off-medication condition
Change from Baseline in the number of steps on the Timed Up and Go test at 6 months | Baseline and 6 months
  in the off-medication condition
Change from Baseline in the Movement Disorder Society-sponsord Unified Parkinson's Disease Rating Scale Part III at 6 months | Baseline and 6 months
  In the off-medication condition, scores could range from 0 (no movement symptoms) to 72 (severe movement symptoms).
Change from Baseline in balance confidence on the Activities-Specific Balance Confidence Scale (ABC) at 12 months | Baseline and 12 months
  The scores could range from 0 (no balance confidence) to 100 (good balance confidence).
Change from Baseline in balance confidence on the Activities-Specific Balance Confidence Scale (ABC) at 6 months | Baseline and 6 months
  The scores could range from 0 (no balance confidence) to 100 (good balance confidence).
Change from Baseline in freezing of gait on the New Freezing of Gait Questionnaire (NFOG-Q) at 12 months | Baseline and 12 months
  The scores could range from 0 (no freezing of gait) to 28 (severe freezing of gait).
Change from Baseline in freezing of gait on the New Freezing of Gait Questionnaire (NFOG-Q) at 6 months | Baseline and 6 months
  The scores could range from 0 (no freezing of gait) to 28 (severe freezing of gait).
Change from Baseline in dysphagia severity on the Swallowing Disturbance Questionnaire (SDQ) at 12 months | Baseline and 12 months
  The scores could range from 0 (no dysphagia) to 44.5 (severe dysphagia).
Change from Baseline in dysphagia severity on the Swallowing Disturbance Questionnaire (SDQ) at 6 months | Baseline and 6 months
  The scores could range from 0 (no dysphagia) to 44.5 (severe dysphagia).
Change from Baseline in gait impairment on the Gait and Fall Questionnaire (GFQ) at 12 months | Baseline and 12 months
  The scores could range from 0 (no gait impairment) to 64 (severe gait impairment).
Change from Baseline in gait impairment on the Gait and Fall Questionnaire (GFQ) at 6 months | Baseline and 6 months
  The scores could range from 0 (no gait impairment) to 64 (severe gait impairment).
Change from Baseline in medication usage on the Levodopa Equivalent Daily Dose at 12 months | Baseline and 12 months
Change from Baseline in medication usage on the Levodopa Equivalent Daily Dose at 6 months | Baseline and 6 months
Change from Baseline in maximal phonatory time at 12 months | Baseline and 12 months
Change from Baseline in maximal phonatory time at 6 months | Baseline and 6 months
Change from Baseline in dysphonia severity index (DSI) at 12 months | Baseline and 12 months
  DSI=0.13 x MPT + 0.0053 x F-High - 0.26 x I-Low - 1.18 x Jitter (%) + 12.4. The DSI for perceptually normal voices equals +5 and for severely dysphonic voices -5. The more negative the patient's index is, the worse is his or her vocal quality.
Change from Baseline in dysphonia severity index (DSI) at 6 months | Baseline and 6 months
  DSI=0.13 x MPT + 0.0053 x F-High - 0.26 x I-Low - 1.18 x Jitter (%) + 12.4. The DSI for perceptually normal voices equals +5 and for severely dysphonic voices -5. The more negative the patient's index is, the worse is his or her vocal quality.
Change from Baseline in cognition on the Montreal Cognitive Assessment at 12 months | Baseline and 12 months
  The scores could range from 0 (severe cognition impairment) to 30 (no cognition impairment).
Change from Baseline in cognition on the Montreal Cognitive Assessment at 6 months | Baseline and 6 months
  The scores could range from 0 (severe cognition impairment) to 30 (no cognition impairment).
Adverse events | up to 12 months after surgery
Change from Baseline in balance ability on the Burg Balance Scale (BBS) at 6 months | Baseline and 6 months
  In the off-medication condition, the scores could range from 0 (severe balance problem) to 56 (no balance problem).
Change from Baseline in the number of freezing episodes on the Timed Up and Go test at 6 months | Baseline and 6 months
  in the off-medication condition

OTHER OUTCOMES:
Change from Baseline in stride length on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in stride length on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in stride velocity on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in stride velocity on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in step length on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in step length on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in step velocity on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in step velocity on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in swing phase/stance phase on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in swing phase/stance phase on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in double support phase on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in double support phase on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in cadence on the Wearable Motion and Gait Quantification System (MATRIX) at 12 months | Baseline and 12 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.
Change from Baseline in cadence on the Wearable Motion and Gait Quantification System (MATRIX) at 6 months | Baseline and 6 months
  In the off-medication condition, the parameters will be recorded by the wearable quantification system during the walking test.

CONTACTS AND LOCATIONS:
Overall Officials: Dianyou Li, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China